CLINICAL TRIAL: NCT02845297
Title: Phase 2 Study of Azacitidine in Combination With Pembrolizumab in Relapsed/Refractory Acute Myeloid Leukemia (AML) Patients and in Newly Diagnosed Older (≥65 Years) AML Patients
Brief Title: Study of Azacitidine in Combination With Pembrolizumab in R/R AML Patients and in Newly Diagnosed Older Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J1651; IRB00098812 (Other: JHM IRB)
Record Dates: First submitted 2016-07-18; First posted 2016-07-27 (Estimated); Results first posted 2023-03-01 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — pembrolizumab; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Safety Run In Phase (only Cohort 1): (Experimental): The treatment of relapsed and refractory AML patients.
  Interventions: Drug: pembrolizumab; Drug: Azacitadine
- Cohort 2 (Experimental): The treatment of newly diagnosed AML patients (≥ 65 years) who are not candidates for intensive induction chemotherapy.
  Interventions: Drug: pembrolizumab; Drug: Azacitadine

INTERVENTIONS:
Drug: pembrolizumab — Intravenous pembrolizumab
  Other Names: MK-3475
Drug: Azacitadine — Intravenous or subcutaneous
  Other Names: Vidaza

SUMMARY:
This is a multicenter, nonrandomized, open-label phase 2 study (with a safety run-in phase) of azacitidine (AZA) 75 mg/m2 given IV or SQ on days 1-7 every 28 days in combination with pembrolizumab 200 mg given IV every 3 weeks (starting on day 8 of cycle 1). The dose/schedule of AZA selected for this study is FDA approved for patients with MDS/AML.

DETAILED DESCRIPTION:
Acute myeloid leukemia (AML) remains a therapeutic challenge. Although 60-80% of newly diagnosed patients with AML respond to induction chemotherapy, the relapse rate remains high (40%-50%) even after allogeneic stem cell transplant (alloHSCT). Data suggests that epigenetic therapy with azacitidine combined with blockade of PD-1/PD-L1 pathway is a rational therapeutic approach both in newly diagnosed older patients and those with relapsed and refractory AML. Furthermore, recent data suggest that the addition of PD-1 blockade (nivolumab) to azacitidine in patients with AML who have previously failed hypomethylating agents may induce responses in up to 20% patients

We plan to examine two AML patient cohorts:

Cohort 1: relapsed/refractory AML. Cohort 2: newly diagnosed AML in older patients (≥65 years) not candidates for induction chemotherapy. Azacitidine and pembrolizumab have distinct mechanisms of action with no common overlapping toxicities; however, as azacitidine and pembrolizumab have not been tested previously in combination in AML patients, we plan to start enrollment with Cohort 1 (a safety run-in phase) and include only relapsed/refractory AML patients excluding those relapsing after allogeneic hematopoietic stem cell transplant (alloHSCT). The primary objective of the run in safety phase would be to determine the safe and tolerable dose/schedule of azacitidine and pembrolizumab in patients with AML. We will perform safety run in phase only in Cohort 1 as Cohort 2 patients would be expected to have a same or better tolerability given that they are not heavily pretreated

ELIGIBILITY:
Inclusion Criteria:

Cohort #1

1. Have histologically or cytologically confirmed relapsed or refractory AML (i.e. ≥5% blasts by manual differential on bone marrow aspirate/biopsy/flow cytometry), excluding acute promyelocytic leukemia (APL; FAB M3; t(15;17))
2. Be willing and able to provide written informed consent/assent for the trial.
3. Be > 18 years of age on day of signing informed consent.
4. Not be appropriate candidate for intensive salvage chemotherapy due to co-morbidities or other disease- or treatment-related factors.

   NOTE: Subjects who received prior treatment with hypomethylating agents either for Myelodysplastic Syndrome (MDS), Myeloproliferative Neoplasm (MPN), or AML will be eligible if they achieved response to hypomethylating agents in the past (PR or CR) and did not progress while receiving therapy with hypomethylating agents.

   NOTE: Subjects who had prior allogeneic stem cell transplant (alloHSCT) will be eligible as long as they have been at least 3 months after allogeneic HSCT and are off of all immune suppression for at least 3 weeks (>21 days) and have no evidence of active graft versus host disease (GVHD). Subjects with prior alloHSCT will NOT be eligible for enrollment during the safety run in phase.
5. Demonstrate adequate organ function as defined in Table 1, all screening labs should be performed within 14 days of treatment initiation.
6. ECOG performance status ≤ 2.
7. A projected life expectancy of at least 12 weeks.
8. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
9. Female subjects of childbearing potential (Section 5.8.2) must be willing to use an adequate method of contraception as outlined in Section 5.8.2 - Contraception, for the course of the study through 120 days after the last dose of study medication.

   Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
10. Male subjects of childbearing potential (Section 5.8.2) must agree to use an adequate method of contraception as outlined in Section 5.8.2- Contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy.

    Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
11. As determined by the enrolling physician or protocol designee, ability of the patient to understand and comply with study procedures for the entire length of the study.

Cohort #2

1. Have histologically and cytologically confirmed newly diagnosed AML (i.e. ≥ 20% blasts by manual differential on bone marrow aspirate/biopsy and/or in peripheral blood), excluding acute promyelocytic leukemia (APL; FAB M3, t (15;17))
2. Be willing and able to provide written informed consent/assent for the trial.
3. Be ≥65 years of age on day of signing informed consent.
4. Have received NO prior treatment for AML with the exception of hydroxyurea/leukapheresis.

   NOTE: Subjects may have been treated for pre-existent myeloid disorder such as Myelodysplastic Syndrome or Myeloproliferative Neoplasm excluding hypomethylating agents.
5. Demonstrate adequate organ function as defined in Table 1, all screening labs should be performed within 14 days of treatment initiation.
6. ECOG performance status ≤ 2.
7. A projected life expectancy of at least 12 weeks.
8. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
9. Female subjects of childbearing potential (Section 5.8.2) must be willing to use an adequate method of contraception as outlined in Section 5.8.2 - Contraception, for the course of the study through 120 days after the last dose of study medication.

   Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
10. Male subjects of childbearing potential (Section 5.8.2) must agree to use an adequate method of contraception as outlined in Section 5.8.2- Contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy.

    Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
11. As determined by the enrolling physician or protocol designee, ability of the patient to understand and comply with study procedures for the entire length of the study.

Adequate Organ Function Laboratory Values

White blood cell (WBC) count <30,000 /mcL

Serum creatinine OR Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤1.5 X upper limit of normal (ULN) OR ≥60 mL/min for subject with creatinine levels > 1.5 X institutional ULN Serum total bilirubin ≤ 1.5 X ULN* AST (SGOT) and ALT (SGPT) ≤ 3 X ULN Albumin >2.5 mg/dL International Normalized Ratio (INR) or Prothrombin Time (PT) Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants

≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants

Exclusion Criteria:

Cohort #1

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.

   NOTE: Subjects who were treated on a clinical study of allogeneic stem cell transplant (alloHSCT) will be eligible if they are at least 3 months after allogeneic HCT and are at least 3 weeks (>21 days) off of all immune suppression and have no evidence of active GVHD (physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency is allowed). Subjects with prior alloHSCT will not be eligible for enrollment during the safety run in phase.
2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
3. Has a known history of active TB (Bacillus Tuberculosis)
4. Hypersensitivity to pembrolizumab or any of its excipients.
5. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
6. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks or growth factors within 1 week prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   * Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
   * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
7. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
8. Has known active central nervous system (CNS) leukemia. Subjects with previously treated CNS leukemia may participate provided that they have documented clearance of CNS leukemia and are not actively treated with intrathecal chemotherapy.
9. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. Subjects that require intermittent use of bronchodilators or local steroid injections will not be excluded from the study.
10. Has known history of, or any evidence of active, non-infectious pneumonitis.
11. Has an active uncontrolled infection requiring systemic therapy (viral, bacterial or fungal). Patients with infection under active treatment and controlled with antibiotics are eligible.
12. Has a white blood cell count > 30 x 109/L. NOTE: Leukapheresis and Hydroxyurea is permitted to meet this criterion and should be stopped ≥12 hours before starting treatment on the study.
13. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
14. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
15. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
16. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
17. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
18. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
19. Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Cohort #2

1. Has received treatment with hypomethylating agent for pre-existent myeloid disorder such Myelodysplastic Syndrome (MDS) or Myeloproliferative Neoplasm (MPN).
2. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment for pre-existent myeloid disorder such as MDS or MPN.
3. Not be eligible for treatment with a standard cytarabine and anthracycline or similar intensive induction chemotherapy due to co-morbidities or other factors, or is unwilling to receive intensive induction therapy.
4. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
5. Has a known history of active TB (Bacillus Tuberculosis)
6. Hypersensitivity to pembrolizumab or any of its excipients.
7. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
8. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks or growth factors within 1 week prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   * Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
   * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
9. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
10. Has known active central nervous system (CNS) leukemia. Subjects with previously treated CNS leukemia may participate provided that they have documented clearance of CNS leukemia and are not actively treated with intrathecal chemotherapy.
11. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. Subjects that require intermittent use of bronchodilators or local steroid injections will not be excluded from the study.
12. Has known history of, or any evidence of active, non-infectious pneumonitis.
13. Has an active uncontrolled infection requiring systemic therapy (viral, bacterial or fungal). Patients with infection under active treatment and controlled with antibiotics are eligible.
14. Has a white blood cell count > 30 x 109/L. NOTE: Leukapheresis and hydroxyurea is permitted to meet this criterion and should be stopped ≥12 hours before starting treatment on the study.
15. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
16. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
17. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
18. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
19. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
20. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
21. Has received a live vaccine within 30 days of planned start of study therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2022-04 (Actual); Study Completion 2022-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ivana Gojo, MD, Principal Investigator — Johns Hopkins University
Locations (3):
- United States (3):
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - University of North Carolina Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Medical University of South Carolina Hollings Cancer Center, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rutella S, Vadakekolathu J, Mazziotta F, Reeder S, Yau TO, Mukhopadhyay R, Dickins B, Altmann H, Kramer M, Knaus HA, Blazar BR, Radojcic V, Zeidner JF, Arruda A, Wang B, Abbas HA, Minden MD, Tasian SK, Bornhauser M, Gojo I, Luznik L. Immune dysfunction signatures predict outcomes and define checkpoint blockade-unresponsive microenvironments in acute myeloid leukemia. J Clin Invest. 2022 Nov 1;132(21):e159579. doi: 10.1172/JCI159579. PMID 36099049

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 40 participants started in phase 1 of the study followed by an additional 27 participants in phase 2
Groups:
- Safety Run in Phase (Only Cohort 1): The treatment of relapsed/refractory AML patients receiving azacitidine and pembrolizumab.
- Cohort 2 (Newly Diagnosed Patients): New diagnosed older patients (greater than or equal to 65 years of age) who are not candidates for intensive induction chemotherapy receiving azacitidine and pembrolizumab.
Period: Phase 1 (2 Years)
Arm/Group | Safety Run in Phase (Only Cohort 1) | Cohort 2 (Newly Diagnosed Patients)
Started | 40 | 0
Completed | 40 | 0
Not Completed | 0 | 0
Period: Phase (2 Years)
Arm/Group | Safety Run in Phase (Only Cohort 1) | Cohort 2 (Newly Diagnosed Patients)
Started | 0 | 27
Completed | 0 | 27
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: Relapsed/Refractory AML Patients: The treatment of relapsed and refractory AML patients.
  pembrolizumab: Intravenous pembrolizumab
  Azacitadine: Intravenous or subcutaneous
- Cohort 2: Newly Diagnosed Older Patients Not Eligible for Intensive Chemo: The treatment of newly diagnosed AML patients (≥ 65 years) who are not candidates for intensive induction chemotherapy.
  pembrolizumab: Intravenous pembrolizumab 200 mg every 3 weeks
  Azacitadine: Intravenous or subcutaneous
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Relapsed/Refractory AML Patients | Cohort 2: Newly Diagnosed Older Patients Not Eligible for Intensive Chemo | Total
Number analyzed (Participants) | 40 | 27 | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 0 | 22
  >=65 years | 18 | 27 | 45
Age, Continuous [Mean (Full Range); unit: years] | 65 [33 to 83] | 75 [69 to 83] | 70 [33 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 3 | 21
  Male | 22 | 24 | 46
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40 | 27 | 67

OUTCOME MEASURES:

1. Primary Outcome: Maximal Tolerable Dose of Pembrolizumab for Cohort 1
Description: The primary objective is to determine the safe and tolerable dose for both the relapsed/refractory AML patients.
Time Frame: 3- 28 day cycles
Population: This outcome was assessed only in Cohort 1.
Measure: Number; unit: mg
Groups:
- Cohort 1: Relapsed/Refractory AML Patients: Relapsed/refractory AML patients.
- Cohort 2: Newly Diagnosed Older Patients Not Eligible for Intensive Chemo: New diagnosed older patients (greater than or equal to 65 years of age) who are not candidates for intensive induction chemotherapy.
Arm/Group | Cohort 1: Relapsed/Refractory AML Patients | Cohort 2: Newly Diagnosed Older Patients Not Eligible for Intensive Chemo
Number analyzed (Participants) | 40 | 0
mg | 200 |

2. Secondary Outcome: Number of Participants Who Had Complete Remission/Complete Remission With Incomplete Recovery
Description: Response will be assessed using the International European LeukemiaNet Guidelines in AML63 and IWG Modified Response Criteria (2006) for CR and CRi. CR is bone marrow blasts <5%; absence of circulating blasts; ANC > or = 1, 000/mcL; platelet count > or = 100,000/mcL. CRi is all CR criteria except for residual neutropenia (<1,000/mcL) or thrombocytopenia (<100,000/mcL).
Time Frame: 3-28 day cycles
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 2: Newly Diagnosed Older Patients Not Eligible for Intensive Chemo: The treatment of newly diagnosed AML patients (≥ 65 years) who are not candidates for intensive induction chemotherapy.
  pembrolizumab: Intravenous pembrolizumab
  Azacitadine: Intravenous or subcutaneous
Arm/Group | Cohort 1: Relapsed/Refractory AML Patients | Cohort 2: Newly Diagnosed Older Patients Not Eligible for Intensive Chemo
Number analyzed (Participants) | 40 | 27
Participants | 5 | 13

ADVERSE EVENTS:
Time Frame: Adverse event data will be collected at the time of participant consent until 30 days from the end of treatment. Serious adverse events will be collected for 90 days after end of treatment. After documented disease progression each subject will be followed by telephone for overall survival until death, withdrawal of consent, or the end of the study, whichever occurs first. Adverse event assessment occurred for up to 2.5 years on average for all patients.
Arm/Group | Cohort 1: Relapsed/Refractory AML Patients | Cohort 2: Newly Diagnosed Older Patients Not Eligible for Intensive Chemo
All-Cause Mortality (participants affected / at risk) | 39/40 | 23/27
Serious Adverse Events (participants affected / at risk) | 4/40 | 1/27
Other Adverse Events (participants affected / at risk) | 6/40 | 0/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Relapsed/Refractory AML Patients (N=40) | Cohort 2: Newly Diagnosed Older Patients Not Eligible for Intensive Chemo (N=27)
Sepsis (Infections and infestations) | 4 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Relapsed/Refractory AML Patients (N=40) | Cohort 2: Newly Diagnosed Older Patients Not Eligible for Intensive Chemo (N=27)
Lung Infection (Infections and infestations) | 6 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-14): https://cdn.clinicaltrials.gov/large-docs/97/NCT02845297/Prot_SAP_000.pdf